CLINICAL TRIAL: NCT01556451
Title: An Open-label, Single-arm, Multi-center, Phase IV Clinical Trial to Evaluate the Safety, Tolerability, and Immunogenicity of ZOSTAVAX™ in Healthy Adults in Korea
Brief Title: ZOSTAVAX™ Safety and Immunogenicity in Korean Adults (V211-034)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V211-034
Record Dates: First submitted 2012-02-17; First posted 2012-03-16 (Estimated); Results first posted 2013-09-23 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-03

CONDITIONS: Herpes Zoster; Shingles
MeSH Terms: conditions — Herpes Zoster | interventions — Herpes Zoster Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Zoster Vaccine Live (Experimental): Single subcutaneous injection of 0.65 mL in the deltoid region of arm on Day 1
  Interventions: Biological: Zoster Vaccine Live

INTERVENTIONS:
Biological: Zoster Vaccine Live — Zoster vaccine live
  Other Names: ZOSTAVAX™; V211

SUMMARY:
This study will evaluate the safety, tolerability, and immunogenicity of ZOSTAVAX™ in Korean adults. Approximately 180 herpes zoster history negative subjects ≥ 50 years of age will be enrolled in the study. Each subject will receive a single dose of ZOSTAVAX™. No statistical hypothesis testing will be conducted in the study.

ELIGIBILITY:
Inclusion Criteria:

* No fever on day of vaccination
* Females have a negative pregnancy test and use an acceptable method of birth control, or are postmenopausal
* Underlying chronic illness must be stable

Exclusion Criteria:

* History of hypersensitivity reaction to any vaccine component
* Prior history of herpes zoster
* Prior receipt of varicella or zoster vaccine
* Pregnant or breastfeeding
* Have recently received immunoglobulins or blood products other than autologous blood transfusion
* Received any inactivated other live virus vaccine within 4 weeks prior to vaccination, or is expected to received any other live virus vaccine during the duration of the study
* Received any inactivated vaccine within 7 days prior to vaccination, or is expected to receive any inactivated vaccine during the duration of the study
* Use of immunosuppressive therapy
* Known or suspected immune dysfunction
* Use of nontopical antiviral therapy with activity against herpes virus
* Known or suspected active untreated tuberculosis

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2012-04; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Choi WS, Choi JH, Choi JY, Eom JS, Kim SI, Pai H, Peck KR, Sohn JW, Cheong HJ. Immunogenicity and Safety of a Live Attenuated Zoster Vaccine (ZOSTAVAX) in Korean Adults. J Korean Med Sci. 2016 Jan;31(1):13-7. doi: 10.3346/jkms.2016.31.1.13. Epub 2015 Dec 24. PMID 26770032

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Zoster Vaccine Live
Started | 180
Completed | 180
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Zoster Vaccine Live
Number analyzed (Participants) | 180
Age, Customized [Number; unit: Participants]
  Between 50 and 59 years | 89
  60 years or older | 91
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 136
  Male | 44

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Fold Rise (GMFR) From Day 1 in Varicella Zoster Virus (VZV) Antibody
Description: Blood samples collected prevaccination on Day 1 and Week 4 postvaccination were analyzed using a glycoprotein enzyme-linked immunosorbent assay (gpELISA) to detect Immunoglobulin G antibody to VZV. The GMFR reports the geometric mean of the ratio of individual participant VZV antibody titers at Week 4 postvaccination / Day 1 (Baseline).
Time Frame: Day 1 (Baseline) and Week 4 postvaccination
Population: The population analyzed included all participants who received Zoster Vaccine Live and were not excluded at the request of the Institutional Review Board and did not have major deviations from the protocol procedures
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Zoster Vaccine Live
Number analyzed (Participants) | 166
Ratio | 2.8 [2.5 to 3.1]

2. Primary Outcome: Geometric Mean Titer (GMT) of VZV Antibody
Description: Blood samples collected prevaccination on Day 1 and Week 4 postvaccination were analyzed using a gpELISA to detect Immunoglobulin G antibody to VZV
Time Frame: Day 1 (Baseline) and 4 weeks postvaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: gpELISA units/mL
Arm/Group | Zoster Vaccine Live
Number analyzed (Participants) | 166
gpELISA units/mL
  Day 1 (Baseline) | 66.9 [59.2 to 75.5]
  Week 4 postvaccination | 185.4 [167.0 to 205.9]

3. Primary Outcome: Percentage of Participants With Clinical Adverse Experiences
Description: An adverse experience was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of study vaccine, whether or not considered related to the use of the product. Any worsening of a preexisting condition which is temporally associated with the use of the study vaccine is also an adverse experience.
Time Frame: Up to 42 days postvaccination
Population: Safety population which included all vaccinated participants who had any safety follow-up
Measure: Number; unit: Percentage of Participants
Arm/Group | Zoster Vaccine Live
Number analyzed (Participants) | 180
Percentage of Participants
  Injection site adverse experiences | 53.3
  Non-injection site adverse experiences | 24.4

4. Primary Outcome: Percentage of Participants Discontinued Due to Clinical Adverse Experiences
Time Frame: Up to 42 days postvaccination
Population: Safety population which included all vaccinated participants who had any safety follow-up
Measure: Number; unit: Percentage of Participants
Arm/Group | Zoster Vaccine Live
Number analyzed (Participants) | 180
Percentage of Participants | 0

ADVERSE EVENTS:
Time Frame: Up to 42 days postvaccination
Arm/Group | Zoster Vaccine Live
Serious Adverse Events (participants affected / at risk) | 3/180
Other Adverse Events (participants affected / at risk) | 96/180
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zoster Vaccine Live (N=180)
Anal Fistula (Gastrointestinal disorders) | 1 (1)
Gastric Polyps (Gastrointestinal disorders) | 1 (1)
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zoster Vaccine Live (N=180)
Injection-Site Erythema (General disorders) | 81 (81)
Injection-Site Pain (General disorders) | 50 (51)
Injection-Site Swelling (General disorders) | 68 (68)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission.